CLINICAL TRIAL: NCT03565549
Title: VAGABOND: a Mnemonic to Aid in the Memory Retention of the Canadian CT Head Rule for Patients With Minor Head Injury: A Randomized Controlled Trial on Interns and Senior Medical Students
Brief Title: VAGABOND: a Mnemonic to Aid in the Memory Retention of the Canadian CT Head Rule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Ammar Al Kashmiri, Senior consultant, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SultanQU
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Traumatic Brain Injury; Education
Keywords: Brain; Trauma; Medical education; Emergency department
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries; Emergencies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mnemonic (Experimental): Intervention group will receive a mnemonic aid to remember the CCHR
  Interventions: Behavioral: Mnemonic
- CCHR rule (Active Comparator): The control group will receive the CCHR only
  Interventions: Behavioral: CCHR rule

INTERVENTIONS:
Behavioral: Mnemonic — A mnemonic used as a memory aid
  Arms: Mnemonic
Behavioral: CCHR rule — A list of the CCHR items
  Arms: CCHR rule

SUMMARY:
The aim of this study is to assess the effectiveness and usefulness of a simple one word mnemonic in the memory retention of the different components of the Canadian CT Head Rule (CCHR) in senior medical students and interns. The CCHR, a clinical decision rule used by emergency physicians to determine the need of head CT in the context of minor traumatic brain injury (mTBI). A rapid recall of the rule in the clinical setting would be expected to improve its utilization and overcome one of the barriers in its implementation. This would ultimately result in better utilization of resources and reduction in unnecessary exposure to radiation.

DETAILED DESCRIPTION:
Introduction

Minor head injury is a serious public health problem. It is defined as a history of loss of consciousness, amnesia, or disorientation and a Glasgow Coma Scale (GCS) score of 13-15 [1]. Patients with minor head injury are frequently encountered in the emergency department and the outpatient settings [2]. In the United States, it is estimated that each year there are about 1.2 million Emergency Department (ED) visits and 800,000 visits to the outpatient setting related to minor head injury [2]. Although most patients with minor head injury can be discharged without sequelae after observation, a small proportion deteriorates and requires neurosurgical intervention for intracranial pathology [3]. Therefore, early diagnosis of such injuries by computed tomography (CT) followed by early surgery is very important in the treatment of those patients. Therefore, when faced with such situation, clinicians have to make the decision whether further investigation in the form of CT imaging of the head is necessary to rule out an intracranial lesion. Not imaging a minor head injury could potentially lead to significant consequences if an intracranial pathology is missed. On the other hand, imaging all patients will lead to unacceptable exposure to ionizing radiation and waste valuable health resources.

Clinical decision rules (CDRs) are tools that attempt to formally test, simplify, and increase the accuracy of clinicians' diagnostic and prognostic assessments. They guide clinicians, establish pretest probability, provide screening tests for common problems, and estimate risk [4]. A number of CDRs have been developed to guide clinicians dealing with minor head injuries on deciding whether CT scan of the head is indicated or not [1,5,6,7,8,9,10,11,12]. Among the multitude of CDRs, the Canadian CT Head Rule (CCHR) has been repeatedly shown to be useful with good sensitivity and specificity [13,14]. It was first developed and tested among 3212 patients with head injuries in 10 Canadian institutions between 1996 and 1999 and published in 2001[1].

The CCHR consists of five high-risk factors (failure to reach GCS of 15 within 2 h, suspected open skull fracture, any sign of basal skull fracture, vomiting ≥2 episodes, or age ≥65 years) and two additional medium-risk factors (amnesia before impact >30 min and dangerous mechanism of injury). The high-risk factors are 100% sensitive for predicting need for neurological intervention, and would require only 32% of patients to undergo CT. The medium-risk factors are 98·4% sensitive and 49·6% specific for predicting clinically important brain injury, and would require only 54% of patients to undergo CT [1].

Despite its demonstrated validity, awareness and use of the rule remains low in many parts of the developed world, including Canada [15]. In fact there is evidence that implementation of the rule did not lead to a reduction in emergency department use of CT imaging and in some occasions there was actually an increase over time in use of CT scans [16]. Several barriers of implementation have been suggested. One of these is physicians' forgetting the details of the rule at the bedside [17]. Having a simple mnemonic that acts as a memory aid to the different components of the rule may help overcome this barrier. Mnemonics have been shown to enhance retention of clinical decision rules such as the Ottawa Ankle and Foot Rules [18]. Therefore, this study proposes the hypothesis that a mnemonic to remember the CCHR will enhance retention of the components of this clinical decision rule by physicians and medical students.

Method:

This is a single-blinded randomized controlled trial to evaluate whether the use of a mnemonic would improve mid-term and long-term knowledge and retention of the CCHR. The participants will be interns and medical students from the Sultan Qaboos University and Oman Medical College. The study tool will be an online survey that will be emailed to all enrolled medical students in both institutions. The initial email will gather demographic and level of education of participants and their initial knowledge about the CCHR. Then participants will be randomized to receive either a table of the rule produced by the developers of the rule listing the CCHR and a second group will receive the mnemonic. The second email will measure the immediate retention of the rule. A follow up email six months after the randomization will assess the retention of the CCHR between the two arms of the study.

The study will aim to recruit all interns and final year medical students. The study will require at least 150 participants in each arm in order to attain 95% power in detecting a 5% difference between variable of the two arms. Randomization will be done using a software program.

The mnemonic VAGABOND will be used to enhance students' retention of the CCHR in this study. The mnemonic stands for:

V for Vomiting more than 2 times A for Amnesia G for GCS less than 15 for more than 2 hours A for Age more than 65 years B for Basal skull fracture ON for OpeN skull fracture D for Dangerous mechanism

The questionnaires are accessible on the following weblinks:

https://docs.google.com/forms/d/1Q3EltuGLuedWJ6w7mzbXi8j4VXCW7vMnq6ThI-rAtVo/edit?ts=5b08ccb1

https://docs.google.com/forms/d/17QbSQEWdqb97Qhlz2hA5gnAIMDcJkHB5bsK8EL4mG5s/edit

Data will be directly entered into a pre-populated Statistical Package for Social Sciences (SPSS) datasheet. The study will present a descriptive analysis of all the variables collected. In order to assess the significance of differences in the variables between the two arms of participants, a series of Chi-Square tests and the Fisher exact tests will be used where appropriate. The Statistical Package for Social Sciences (SPSS) software will be utilized in the data analysis

Implications:

The study will assess whether the use of a mnemonic enhances the awareness of a clinical decision rule among interns and medical students. It will highlight the value of using simple mnemonics in teaching clinical decision-making. Such data is valuable for medical educators in other settings where critical clinical decisions can be made based on available rules.

ELIGIBILITY:
Inclusion Criteria:

* all final year medical students and interns

Exclusion Criteria:

* none

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
memory retention of the Canadian CT Head Rule | 6 months
  the effectiveness and usefulness of a simple one word mnemonic in the memory retention of the different components of the Canadian CT Head Rule

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Qaboos University, Muscat, Oman